CLINICAL TRIAL: NCT02852798
Title: Clinical Study of Apatinib Mesylate Tablets Combined With Docetaxel Monotherapy as Second-line Therapy of Advanced EGFR Wild-type, Non-squamous, Non-small-cell Lung Cancer
Brief Title: Apatinib Combined With Docetaxel Monotherapy as Second-line Therapy of Advanced EGFR WT, Non-squamous NSCLC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jiangsu ShengDiYa Medicine Co., Ltd. (Other)
Collaborators: Dongguan People's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: HRSZ201608
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Nonsquamous Nonsmall Cell Neoplasm of Lung
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Apatinib Combined With Docetaxel — Docetaxel 75 mg/ (m2.d)IV gtt 1h d1 q3w Apatinib Mesylate Tablets : 500 mg qd, 4 weeks as one cycle for continuous drug administration
  Other Names: AITAN

SUMMARY:
This is a clinical study of Apatinib Mesylate Tablets combined with docetaxel monotherapy as second-line therapy of advanced EGFR wild-type, non-squamous, non-small-cell lung cancer.

DETAILED DESCRIPTION:
In order to seek high-efficiency, low-toxicity anti-angiogenic drugs, Jiangsu Hengrui Medical Co., Ltd has developed an efficient VEGFR2 tyrosine kinase inhibitor (TKI) - Apatinib. This drug works mainly by inhibiting VEGFR2 to produce the anti-angiogenic effects and treat malignant tumors. Apatinib was shown to have good tumor growth-inhibiting activity against lung cancer in both in vivo and in vitro experiments.

This study aims to further validate the efficacy and safety of Apatinib combined with chemotherapeutics in the treatment of advanced EGFR wild-type non-squamous, non-small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old
* Pathologically Confirmed advanced (stage IIIB, and IV) non-squamous, non-small cell lung cancer, with measurable lesions (long diameter of tumor lesion according to CT scanning ≥10 mm, short diameter of lymph nodes according to CT scanning ≥15 mm, thickness according to CT scanning no more than 5 mm, measurable lesions which have not been treated with radiotherapy, cryotherapy or other local treatment)
* EGFR mutation detection confirmed EGFR mutation negative (EGFR wild-type)
* The patients have completed at least 2 cycles of first-line combined chemotherapy (including a platinum-based chemotherapy, 2-week or 3-week regimen). Efficacy evaluation indicates PD. No more than 28 days has passed since the last chemotherapy cycle. Patients who previously received treatment with EGFR-TKI could be included
* ECOG Score: 0-3
* Expected survival period ≥ 3 months
* The damages caused by other treatments have been recovered (NCI-CTCAE version 4.0 grading ≤ grade 1), the interval for administration of nitrourea or mitomycin ≥ 6 weeks, or administration of other cytotoxic drugs bevacizumab (Avastin), radiotherapy or surgery ≥ 4 weeks, or administration of EGFR TKI molecular target drugs ≥ 2 weeks
* Functions of major organs are normal, i.e. the following criteria should be met:

  1. Routine blood test results meet the criteria (no blood transfusion or use of blood products, and no use of G-CSF or other hematopoietic stimulating factors within 14 days)

     1. HB≥90 g/L
     2. ANC≥15×10^9/L
     3. PLT≥80×10^9/L
  2. The following criteria should be met in the biochemical tests:

     1. TBIL<1.5×ULN
     2. ALT and AST<2.5×ULN;for patients with liver metastasis, ALT and AST >5×ULN
     3. Serum Cr≤1.25×ULN or Endogenous creatinine clearance rate>45 ml/min (Cockcroft-Gault formula)
* Women of childbearing age should have taken reliable contraceptive measures, or received pregnancy test (serum or urine) with a negative result within 7 days before being included, and are willing to take appropriate contraceptive measures during the trial and within 8 weeks after last dose of the study drug. Males who have not received sterilization operation should agree to take appropriate contraceptive measures during the trial and within 8 weeks after last dose of the study drug
* The subjects are voluntary to join this study. They have signed the Informed Consent Form and are willing to coordinate with the follow-up with good compliance.

Exclusion Criteria:

* Patients with quamous carcinoma (including adenosquamous carcinoma ); small cell lung cancer (including small cell cancer and non-small cell mixed lung cancer)
* Patients with active brain metastasis, carcinomatous meningitis, or spinal compression, or disease of brain or pia mater according to the screening test, imaging, CT or MRI tests (patients who have completed the treatment and in a stable condition 21 days before screening could be included, but brain MRI, CT or venography is required to confirm that there are no brain hemorrhage symptoms)
* Imaging (CT or MRI) results indicate that the distance between the tumor and the large vessel ≤ 5 mm, or the existence of central tumors locally invading the large vessel could be detected
* Imaging (CT or MRI) indicates apparent pulmonary cavity or necrotizing tumors.
* Hypertension out of control (systolic pressure≥140 mmHg or diastolic pressure≥90 mmHg, despite optimal drug therapy)
* Patients with myocardial ischemia or myocardial infarction above grade II, or arrhythmia out of control (including QTc interval ≥450 ms for males and ≥470 ms for females)
* Patients with cardiac insufficiency grade III~IV according to NYHA standard, or cardiac color ultrasound indicated LVEF <50%
* Abnormal blood coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds, or APTT >1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment
* Patients treated with anticoagulation agents or Vitamin K antagonist such as Warfarin, heparin, or other similar drugs
* Patients who had obvious hemoptysis within 2 months before screening, or experienced daily hemoptysis with a volume more than half a tea spoon (2.5ml) or above
* Patients who experienced bleeding symptoms of clinical significance within 3 months before screening, or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc
* Patients who manifested arterial/venous thrombus events, e.g. cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism, etc., within 12 months before screening
* Known genetic or acquired bleeding or bleeding tendency (such as hemophilia, blood coagulation dysfunction, thrombocytopenia, and hypersplenism, etc.)
* Patients who have unhealed wounds or fractures for a long time
* Patients who received major surgical operations or experienced severe traumatic injuries, bone fracture, or ulcers within 4 weeks before screening
* Patients with obvious factors affecting absorption of oral drugs, such as difficulties in swallowing, chronic diarrhea and intestinal obstruction, etc
* Occurrence of abdominal fistula, gastrointestinal perforation, or intraperitoneal abscess within 6 months before screening
* Patients whose routine urine tests indicate that urine protein ≥ ++ or verifies that the 24-h urine protein quantitation ≥ 1.0 g
* Patients with clinical symptoms, or dropsy of serous cavity requiring surgical treatment (including hydrothorax, ascites, and hydropericardium)
* Patients who have a history of psychotropic drug abuse and are unable to break the habit, or who have a psychogeny
* Patients who have taken part in other drug clinical tests within 4 weeks before screening
* Confirmed ALK genetic abnormality (gene fusion or mutation)
* Patients who formerly suffered from or currently are complicated with other uncured malignant tumors, except basal cell carcinoma, carcinoma in situ of cervix and superficial bladder cancer that have been cured
* Patients who received the treatment with potent CYP3A4 inhibitors within 7 days before screening, or potent CYP3A4 inducers within 12 days before being included
* Pregnant or lactating women, fertile patients who are unwilling or unable to take effective contraceptive measures
* Conditions determined by investigators to possibly affect the clinical study or determination of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced EGFR wild-type, non-squamous, non-small-cell lung cancer
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year

SECONDARY OUTCOMES:
Overall survival | 1 year
duration of response | 1 year
disease control rate | 1 year
objective remission rate | 1 year

IPD SHARING:
Plan to Share IPD: Undecided